CLINICAL TRIAL: NCT03612661
Title: Piloting a Novel Intuitive Eating Intervention for College Women With Disordered Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20012263
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Disordered Eating Behaviors
Keywords: disordered eating, body image, intuitive eating, undergraduates, college, unhealthy weight control behaviors, eating disorders, weight stigma, weight bias
MeSH Terms: conditions — Disordered Eating Behavior; Feeding and Eating Disorders; Weight Prejudice

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a group or guided self-help condition, of the same intervention, intuitive eating, of the same duration (8 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intuitive Eating Group Intervention (Experimental): Intuitive eating intervention delivered in a group format with 8-10 women, led by 2 facilitators.
  Interventions: Behavioral: Group Intervention
- Intuitive Eating Guided Self-Help (Experimental): Participants in this condition engage in 8 weeks of self-study of the intuitive eating intervention have ~20 minute weekly phone call with a study interventionist.
  Interventions: Behavioral: Guided Self-Help

INTERVENTIONS:
Behavioral: Group Intervention — Participants in the group intervention will attend eight weekly, 90-minute sessions involving group activities and discussions. They will complete homework between sessions to reinforce learning. The intervention focuses on cultivating attunement to bodily sensations and fostering self-compassion to improve physical and mental health.
  Arms: Intuitive Eating Group Intervention
Behavioral: Guided Self-Help — Participants in the GSH condition will follow the intuitive eating content through self-guided study, with eight weekly scheduled phone calls with an interventionist (~20 minutes each). Interventionists will review homework assignments, answer questions, and reinforce adherence. The intervention materials are the same as the group and also focus on cultivating attunement to bodily sensations and fostering self-compassion to improve physical and mental health.
  Arms: Intuitive Eating Guided Self-Help

SUMMARY:
The purpose of this research study is to pilot test a new intervention that helps young adult women learn adaptive eating and exercise strategies, increase their body acceptance, decrease unhealthy weight control behaviors and prevent future eating and problems. This intervention is experimental, and the study will test its feasibility, acceptability, and effectiveness.

DETAILED DESCRIPTION:
The intervention, Intuitive Eating, is an eating approach that addresses important risk factors and promotes adaptive eating attitudes and behaviors. It has three central tenets: 1) unconditional permission to eat when hungry, 2) eating for physical rather than emotional reasons, and 3) eating according to hunger and satiety cues. Intuitive Eating has ten principles that focus on rejecting the dieting mentality, honoring hunger cues, decreasing restrictive behaviors that lead to deprivation and bingeing, challenging rigid food rules, increasing awareness of satiety, discovering the satisfaction of food, coping with emotions without food, respecting and accepting one's body, using exercise as self-care, and balancing nutrition with satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant
* Enrolled in postsecondary education at VCU
* Have body image or eating concerns

Exclusion Criteria:

* Eating disorder threshold risk
* Men
* Pregnant women

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Change in diagnostic eating disorder symptoms | Baseline to 16 weeks
  The Eating Disorder Diagnostic Scale (EDDS) is a brief self-report measure that screens for the presence of subthreshold or threshold levels of ED symptoms. It yields a symptom composite score, to be used as the primary outcome measure. Items assessing body dissatisfaction, overvaluation of shape/weight, and impairment are measured on a 0 to 6-point scale with higher ratings indicating greater body dissatisfaction. Items evaluating the presence of compensatory behaviors and binge eating are rated yes/no and participants indicate the frequency these behaviors have occurred in the prior 3 months.
Change in global eating disorder symptoms | Baseline to 16 weeks
  The EDE-Q is a 28-item self-report version of the Eating Disorder Examination that measures frequency of disordered eating cognitions and behaviors experienced in the previous 28 days. Participants rate the number of days behaviors have occurred in the last 28 days, with 0 = no days and 6 = every day. Yes/no questions identify the presence of compensatory and binge behaviors and participants indicate the frequency of these behaviors over the last 28 days. Higher EDE-Q scores indicate greater eating pathology.
Changes in intuitive eating | Baseline to 16 weeks
  The Intuitive Eating Scale-2 (IES-2) is a 23-item self-report measure of intuitive eating with three subscales: Unconditional Permission to Eat, Eating for Physical Rather Than Emotional Reasons, and Reliance on Hunger and Satiety Cues. Items are rated on a 1 to 5-point scale with higher scores indicating higher levels of intuitive eating.

SECONDARY OUTCOMES:
Change in body appreciation | Baseline to 16 weeks
  The Body Appreciation Scale-2 (BAS-2) is a 10-item measure of positive body image. Specifically, it assesses body appreciation, which reflects acceptance of and favorable opinions and respect towards one's body and a rejection of the narrow beauty ideals promoted through mass media. Items are rated on a 5-point scale with higher scores indicating greater body appreciation.
Changes in dietary restraint | Baseline to 16 weeks
  The Dutch Restrained Eating Scale (DRES) contains 10 items that measure dietary restraint for the purpose of weight loss. Items are rated on a 5-point scale with higher scores reflecting greater dietary restraint.
Changes in body functionality appreciation | Baseline to 16 weeks
  The Functionality Appreciation Scale (FAS) is a 7-item scale that measures appreciation for the functionality of one's body, which is believed to help offset appearance concerns. Items are rated on a 5-point scale with higher scores reflecting greater appreciation for the functionality of one's body.
Changes in interoceptive awareness | Baseline to 16 weeks
  The Interoceptive Awareness subscale of the EDI-3 has 10 items that measure an individual's attunement to their internal state, including perceptions of emotions, hunger, and satiety. Items are rated on a 6-point scale, with higher scores reflecting greater deficits in interoceptive awareness.
Changes in intuitive exercise | Baseline to 16 weeks
  The Intuitive Exercise Scale (IEXS) measures adaptive exercise behaviors that are guided by physical cues and flexibility rather than rigid rules or feelings of obligation. Items are rated on a 5-point scale, with higher scores reflecting more intuitive exercise behaviors.
Changes in weight bias internalization | Baseline to 16 weeks
  The Modified Weight Bias Internalization Scale (WBIS-M) is a modified version of the Weight Bias Internalization Scale that was adapted for use with individuals across the weight spectrum. The WBIS-M measures the degree to which individuals apply weight-based stereotypes to themselves and use those to guide their weight self-evaluations. Items are rated on a 7-point scale, with higher scores reflecting greater degrees of weight bias internalization.
Changes in satisfaction with life | Baseline to 16 weeks
  The Satisfaction with Life Scale (SWLS) is a 5-item scale that assesses global life satisfaction. Items are scored on a 7-point scale, with higher scores reflecting greater life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Mazzeo, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be available by researcher request only after study completion. Interested researchers can email the primary study contact.

DOCUMENTS (1):
  • Informed Consent Form (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03612661/ICF_000.pdf